CLINICAL TRIAL: NCT01959906
Title: Prognostic Value of a Circumferential Section Pane Less Than 1 mm in Esophagectomy for Esophageal Cancer.
Brief Title: Circumferential Section Pane Less Than 1 mm in Esophagectomy for Esophageal Cancer.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Johnny Moons, Datameanager Thoracic Surgery, University Hospital, Gasthuisberg
Other Study IDs: CRM<1mm
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Esophageal Cancer
Keywords: Esophagectomy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- R0: Complete resection
- R1: Incomplete resection, microscopical tumor residu left behind
- CRM<1mm: complete resection (R0), however tumor spreads till less than 1 mm from the section pane.

SUMMARY:
A suspicious circumferential resection margin (CRM), defined as tumor cells within 1 mm of the CRM, is still controversial. The aim of this study was to compare the clinical significance of a suspicious CRM to histologically positive (R1) and negative margin (R0) resections in patients with pT3 esophageal and GE-Junction tumors.

DETAILED DESCRIPTION:
From our prospectively build database 923 consecutive pT3 patients operated between january 1990 and june 2013 were selected. CRM status in patients treated by surgery only (n = 747) or after neoadjuvant therapy (n = 176) was recorded prospectively after surgery.

Kaplan-Meier survival curves were generated, and factors affecting survival were assessed by Cox regression multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* pathologic T3 tumours of esophagus or GEJ

Exclusion Criteria:

* pT other than pT3
* R2 resections

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 923 consecutive pT3 patients operated between january 1990 and june 2013
Sampling Method: Non-Probability Sample
Enrollment: 923 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years after esophagectomy
  5 years overall survival after esophagectomy

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Nafteux, MD, Study Director — University Hospital Leuven, dept. Thoracic Surgery; Katrien Van de Steen, MSc, Principal Investigator — Katholic University Leuven
Locations (1):
- University Hospital Leuven, Leuven, Belgium